CLINICAL TRIAL: NCT00634374
Title: Efficacy of the Rx Medibottle Compared to the Oral Syringe in Delivering Infant-Acceptable Liquid Medication Completely and Accurately: a Controlled Clinical Trial
Brief Title: Administration of a Bitter-Tasting Medication: Comparison Between the Rx Medibottle and the Oral Syringe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Responsible Party: Dr. M Purswani and Dr. J Radhakrishnan, Bronx-Lebanon Hospital Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 09090405
Record Dates: First submitted 2008-02-25; First posted 2008-03-13 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-03

CONDITIONS: Infant Acceptance of Medication
Keywords: Rx medibottle; Oral syringe; Liquid medication; Bitter-tasting; Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Oral Syringe
- 2 (Active Comparator): Rx medibottle
  Interventions: Device: Rx Medibottle

INTERVENTIONS:
Device: Rx Medibottle — Comparing use of the Rx medibottle to the oral syringe in delivering a one-time dose of prednisolone syrup
  Arms: 2

SUMMARY:
Hypothesis: The Rx medibottle is more effective than the oral syringe when giving infants less than 2 years of age a bitter-tasting medication (prednisolone syrup).

Summary: Infants who were admitted to the pediatric floor with a respiratory illness at the Bronx-Lebanon Hospital were offered the chance to take part in the study. If these children needed prednisolone syrup for their treatment, were less than 2 years old and were bottle-fed, and were in stable condition, they qualified. They were randomly assigned (just by chance), into a control arm, where they received medication using the oral syringe, or an intervention arm, where they were given medication using the Rx medibottle. How well the infant accepted the bitter-tasting medication was compared between the two arms using an infant medication acceptance scale. The scale was administered and a score generated by two raters: the nurse who administered the medication, and a child life therapist who witnessed the administration. The time needed to give the medication, the drug delivery device's ability to administer the entire dose of medication and the mother's satisfaction with the method used were also compared between the two arms.

DETAILED DESCRIPTION:
The ability to deliver drugs to infants and children safely and accurately has long been of concern to pediatricians and caregivers. Calibrated oral syringes are accurate in measuring and delivering the required dose, have minimal potential for spillage and are considered the standard drug delivery system for this population. However, infant acceptance of the syringe may not always be favorable. The objective of this study was to compare the Rx medibottle to the oral syringe when used to administer liquid medication to infants. It is a prospective, controlled trial that enrolled infants <2 years of age admitted to a community hospital in the Bronx, who were prescribed a daily dose of 2 mg/kg of prednisolone syrup (15 mg/5 ml) for a respiratory illness. Participants were randomly assigned to receive one dose of prednisolone syrup using the Rx medibottle (intervention arm) or the oral syringe (control arm). The infant medication acceptance scale (MAS) used to evaluate acceptance by the infants was developed and validated by Donna Kraus, Leslie Stohlmeyer and Patricia Hannon and published in the American Journal of Health-System Pharmacy (1999;16:1094-1101).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the pediatric inpatient unit
* Stable condition
* Bottle fed
* Less than 2 years
* Receiving prednisolone syrup (15 mg/5 ml)

Exclusion Criteria:

* Breast fed
* Greater than 2 years

Ages: 2 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Infant acceptance of the bitter-tasting oral liquid medication | On the day of enrollment, with use of drug delivery device

SECONDARY OUTCOMES:
Time needed to administer medication using the drug delivery method | Measured at the time of drug administration by stopwatch
Maternal satisfaction with drug delivery method | At the time of administration or on viewing a videotape of administration
Administration of the entire dose of medication with each drug delivery method | On the day of enrollment, with use of drug delivery device

CONTACTS AND LOCATIONS:
Overall Officials: Murli U Purswani, MD, Principal Investigator — Bronx-Lebanon Hospital Center
Locations (1):
- Bronx-Lebanon Hospital Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Purswani MU, Radhakrishnan J, Irfan KR, Walter-Glickman C, Hagmann S, Neugebauer R. Infant acceptance of a bitter-tasting liquid medication: a randomized controlled trial comparing the Rx Medibottle with an oral syringe. Arch Pediatr Adolesc Med. 2009 Feb;163(2):186-8. doi: 10.1001/archpediatrics.2008.541. PMID 19188654